CLINICAL TRIAL: NCT01466842
Title: Ablation as First Line Treatment in Paroxysmal Atrial Fibrillation
Acronym: AFLIT-PAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AFLIT-PAF 1.2
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (2):
- Catheter ablation (Other)
  Interventions: Procedure: Catheter ablation using cryothermia
- Antiarrhythmic drugs (No Intervention): Three months before starting antiarrhythmic drugs, a subcutaneous loop recorder will be implanted.

INTERVENTIONS:
Procedure: Catheter ablation using cryothermia — Three months before the catheter ablation procedure, a subcutaneous loop recorder will be implanted. The ablation procedure will be performed using cryothermia.
  Arms: Catheter ablation

SUMMARY:
The purpose of this study is to determine whether catheter ablation is more effective than antiarrhythmic drugs in the early stages of paroxysmal atrial fibrillation. In all the patients a subcutaneous loop recorder will be implanted.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* At least three episodes of paroxysmal atrial fibrillation documented on an electrocardiogram or event recording during the last three years
* Never taken antiarrhythmic drugs or at most a pill in the pocket approach
* Willingness, ability and commitment to participate in baseline and follow-up evaluations

Exclusion Criteria:

* Paroxysmal AF for more than three years
* An episode of atrial fibrillation that lasted more than seven days within the past six months
* Persistent/permanent atrial fibrillation
* Atrial fibrillation from reversible cause (i.e. surgery, hyperthyroidism, pericarditis)
* Documented atrial flutter
* Structural heart disease of clinical significance including:

  * Cardiac surgery within six months of screening
  * Unstable symptoms of congestive heart failure (CHF) including NYHA Class III or IV CHF at screening and/or ejection fraction <30% as measured by echocardiography or catheterization
  * Unstable angina
  * Myocardial infarction within six months of screening
  * Surgically corrected atrial septal defect with a patch or closure device
  * LA size > 40mm
* Any prior ablation of the pulmonary veins
* Enrollment in any other ongoing protocol
* Untreatable allergy to contrast media
* Pregnancy
* Any contraindication to cardiac catheterization
* Prosthetic mitral heart valve
* Poor general health that, in the opinion of the Investigator, will not allow the patient to be a good study candidate (i.e. other disease processes, mental capacity, etc.)
* Contraindication to coumadin or heparin
* History of pulmonary embolus or stroke within one year of screening
* Acute pulmonary edema
* Atrial clot on TEE regardless of the patient's anticoagulation medication status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
any recurrence of symptomatic AF or asymptomatic AF and atrial flutter/tachycardia in the absence of AAD therapy during a follow-up period of 6 months | 6 months

SECONDARY OUTCOMES:
any recurrence of symptomatic AF or asymptomatic AF and atrial flutter/tachycardia in the absence of AAD therapy after the initial six months follow-up | 3 years
comparison of the subjective findings of recurrence of AF by the patient through QoL and symptom questionnaires | 3, 6, 12, 24 and 36 months
number of track complications, both acute (during the procedure) and chronic throughout the trial | 3 years
hospitalization rate during a two and a half year follow-up following the initial six months follow-up | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands